CLINICAL TRIAL: NCT07264361
Title: Evaluation of the Safety and Efficacy of the D.D.C Dual-control Technology Spectacle Lenses in Delaying the Progression of Myopia: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: Guangzhou Youyan Vision Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025KYPJ105
Record Dates: First submitted 2025-11-18; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-08

CONDITIONS: Myopia, Progressive
Keywords: Defocus diffusion composite technology; Myopia control
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): D.D.C dual-control technology spectacle lenses
  Interventions: Device: D.D.C dual-control technology spcetacle lenses
- Control (Experimental): Aspheric single-vision spectacle lenes
  Interventions: Device: Aspheric single-vision lenses

INTERVENTIONS:
Device: D.D.C dual-control technology spcetacle lenses — The children in the intervention group will wear D.D.C dual-control technology spcetacle lenses type A for one year, with follow-up visits at baseline, 1 month, 6 months, and 12 months. And then they will be randomized in a 1:1 ratio to either continue with type A lenses or switch to type B lenses, which differ only in the defocus zone. Follow-up visits will be conducted at 13, 18, and 24 months.
  Arms: Intervention
Device: Aspheric single-vision lenses — The children in control group will wear aspheric single-vision lenses for one year, with follow-up visits at baseline, 1 month, 6 months, and 12 months. And then they will be randomized in a 1:1 ratio to either D.D.C dual-control technology spcetacle lenses type A lenses or alternate quarterly (every 3 months) between D.D.C dual-control technology spcetacle lenses type A and type B lenses. Follow-up visits will be conducted at 13, 18, and 24 months.
  Arms: Control

SUMMARY:
The burden of myopia among Chinese children and adolescents is severe and trending toward younger ages, making control of myopia progression a public health priority. Current mainstream strategies include optical interventions, pharmacologic therapy, and environmental measures. Among these strategies, spectacle designs based on optical defocus-such as defocus-incorporated multiple-segment (DIMS) lenses-have demonstrated efficacy; however, the effect of such designs may attenuate over time because of "defocus adaptation." To address this limitation, D.D.C dual-control spectacles employ a densely staggered microlens layout, a gradient-defocus architecture, and an added peripheral "fogging zone" to disrupt the spatial distribution of defocus cues and reduce contrast, thereby delaying adaptation and enhancing myopia-control efficacy.

The present study therefore proposes a 24-month prospective randomized controlled trial in Guangzhou, enrolling eligible myopic adolescents. The trial will first compare 12-month outcomes between D.D.C-A lenses and single-vision lenses, followed by a crossover and alternating-wear phase, to systematically evaluate the safety and efficacy of the D.D.C technology in slowing myopia progression.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 14 years;
* Cycloplegic spherical equivalent refraction between -1.50 D and -5.00 D with astigmatism ≥ -1.50 D in both eyes;
* Absolute interocular difference in spherical equivalent refraction ≤ 1.50 D;
* Binocular best-corrected visual acuity ≥ 1.0;
* Intraocular pressure between 10 and 21 mmHg in both eyes;
* Volunteer to participate in this clinical trial with signature of the informed consent form.

Exclusion Criteria:

* History of eye injury or intraocular surgery or ocular trauma;
* Clinically abnormal slit-lamp findings;
* Abnormal fundus examination;
* Presence of ocular diseases such as cataract, glaucoma, fundus pathology, ocular trauma, manifest strabismus, or any other condition affecting visual function;
* Systemic diseases causing low immunity (such as diabetes, Down's syndrome, rheumatoid arthritis, psychotic patients or other diseases that researchers think are not suitable for wearing glasses);
* Participation in a drug clinical trial within 3 months or a device clinical trial within 1 month prior to enrollment;
* Participation in any myopia control clinical trial within the past 3 months and a history of myopia control interventions (e.g., orthokeratology, atropine);
* Only one eye meeting the inclusion criteria;
* Inability to attend regular ophthalmic examinations.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 316 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in spherical equivalent refraction (SER) from baseline to the 1-year follow-up | Baseline to 1 year
  Change in cycloplegic SER (Diopter) from baseline to 12 months.

SECONDARY OUTCOMES:
Changes in axial length (AL) during the 1-year follow-up | Baseline to 1 year
  Changes in AL (mm) from baseline to 1, 6, and 12 months. AL will be measured using the IOLMaster 700 before cycloplegia.
Changes in spherical equivalent refraction (SER) from baseline during the 1-year follow-up, excluding the 12-month time point. | Baseline to 1 year
  Change in cycloplegic SER (Diopter) from baseline to 1 and 6 months.
Changes in corneal curvature during the 1-year follow-up | Baseline to 1 year
  Changes in corneal curvature (mm) from baseline to 1, 6, and 12 months. Corneal curvature will be measured by IOL Master-700 before cycloplegia.
Changes in anterior chamber depth (ACD) during the 1-year follow-up | Baseline to 1 year
  Changes in ACD (mm) from baseline to 1, 6, and 12 months. ACD will be measured by IOL Master-700 before cycloplegia.
Changes in lens thickness (LT) during the 1-year follow-up | Baseline to 1 year
  Changes in LT (mm) from baseline to 1, 6, and 12 months. LT will be measured by IOL Master-700 before cycloplegia.
Changes in spherical equivalent refraction (SER) at all time points from the 12-month follow-up during the 12-24 month follow-up period | 1 year to 2 years
  Changes in cyclopegic SER (Diopter) from 12 months to 13, 18, and 24 months.
Changes in axial length (AL) from the 12-month follow-up during the 12-24 month follow-up period | 1 year to 2 years
  Changes in AL (mm) from 12 months to 13, 18, and 24 months. AL will be measured using the IOL Master 700 before cyclopegia.
Changes in corneal curvature from the 12-month follow-up during the 12-24 month follow-up period | 1 year to 2 years
  Changes in corneal curvature (mm) from 12 months to 13, 18, and 24 months. Corneal curvature will be measured by IOL Master-700 before cyclopegia.
Changes in anterior chamber depth (ACD) from the 12-month follow-up during the 12-24 month follow-up period | 1 year to 2 years
  Changes in ACD (mm) from 12 months to 13, 18, and 24 months. ACD will be measured by IOL Master-700 before cyclopegia.
Changes in lens thickness (LT) from the 12-month follow-up during the 12-24 month follow-up period | 1 year to 2 years
  Changes in LT (mm) from 12 months to 13, 18, and 24 months. LT will be measured by IOL Master-700 before cyclopegia.
Change in choroidal thickness from baseline to the 1-month follow-up | Baseline to 1 month
  Change in choroidal thickness (μm) from baseline to 1 months.
Change in choroidal thickness from the 12-month to the 13-month follow-up | 1 year to 13 months
  Change in choroidal thickness (μm) from the 12 months to the 13 months.
The proportion of participants who experienced clinically significant myopia progression | Baseline to 2 years
  The proportion of participants who experienced clinically significant myopia progression (>0.5D/year) during the two-year follow-up
Spectacle wear compliance | Baseline to 2 years
  Spectacle wearing time, assessed at each follow-up visit.
The visual scale score during the 2-year follow-up | Baseline to 2 years
  Visual scale score measured by the Chinese version of the pediatric refractive error profile 2 (PREP2) and is scaled from 0 (poor quality of life) to 100 (good quality of life)
The best corrected visual acuity (BCVA) during the 2-year follow-up | Baseline to 2 years
  BCVA will be measured by EDTRS visual acuity chart.
The subjective perception score during the 2-year follow-up | Baseline to 2 years
  Subjective perception score will be measured by questionnaire to test the comfort of wearing spectacles.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Ge, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Greenwald SH, Kuchenbecker JA, Rowlan JS, Neitz J, Neitz M. Role of a Dual Splicing and Amino Acid Code in Myopia, Cone Dysfunction and Cone Dystrophy Associated with L/M Opsin Interchange Mutations. Transl Vis Sci Technol. 2017 May 10;6(3):2. doi: 10.1167/tvst.6.3.2. eCollection 2017 May. PMID 28516000
- [Result] Gupta V, Saxena R, Dhiman R, Phuljhele S, Sharma N. Comparative evaluation of different (peripheral defocus based) spectacle designs in preventing myopia progression: A double-blinded randomised clinical trial. Ophthalmic Physiol Opt. 2025 Sep;45(6):1505-1511. doi: 10.1111/opo.13548. Epub 2025 Jun 24. PMID 40552434
- [Result] Wang M, Ma R, Kuang L, Chen X, Vincent SJ, Tan H, Lai Z, Xu S, Hu Y, Han M, Chen Q, Wang Z, Li L, Yang X. Myopia Control Efficacy of Asymmetric Multipoint Defocus Technique Spectacle Lenses: One-Year Double-Masked Randomized Controlled Trial. Ophthalmology. 2025 Sep;132(9):972-979. doi: 10.1016/j.ophtha.2025.04.022. Epub 2025 Apr 28. PMID 40306584
- [Result] Bao J, Huang Y, Li X, Yang A, Zhou F, Wu J, Wang C, Li Y, Lim EW, Spiegel DP, Drobe B, Chen H. Spectacle Lenses With Aspherical Lenslets for Myopia Control vs Single-Vision Spectacle Lenses: A Randomized Clinical Trial. JAMA Ophthalmol. 2022 May 1;140(5):472-478. doi: 10.1001/jamaophthalmol.2022.0401. PMID 35357402
- [Result] Lam CSY, Tang WC, Tse DY, Lee RPK, Chun RKM, Hasegawa K, Qi H, Hatanaka T, To CH. Defocus Incorporated Multiple Segments (DIMS) spectacle lenses slow myopia progression: a 2-year randomised clinical trial. Br J Ophthalmol. 2020 Mar;104(3):363-368. doi: 10.1136/bjophthalmol-2018-313739. Epub 2019 May 29. PMID 31142465
- [Result] Bullimore MA, Saunders KJ, Baraas RC, Berntsen DA, Chen Z, Chia AWL, Goto S, Jiang J, Lan W, Logan NS, Najjar RP, Polling JR, Read SA, Woodman-Pieterse EC, Szell N, Verkicharla PK, Wu PC, Zhu X, Loughman J, Nagra M, Phillips JR, Tran HDM, Vera-Diaz FA, Yam J, Liu YM, Singh SE, Wildsoet CF. IMI-Interventions for Controlling Myopia Onset and Progression 2025. Invest Ophthalmol Vis Sci. 2025 Sep 2;66(12):39. doi: 10.1167/iovs.66.12.39. PMID 40960225
- [Result] Hu Y, Ding X, Guo X, Chen Y, Zhang J, He M. Association of Age at Myopia Onset With Risk of High Myopia in Adulthood in a 12-Year Follow-up of a Chinese Cohort. JAMA Ophthalmol. 2020 Nov 1;138(11):1129-1134. doi: 10.1001/jamaophthalmol.2020.3451. PMID 32940622
- [Result] Chen Z, Gu D, Wang B, Kang P, Watt K, Yang Z, Zhou X. Significant myopic shift over time: Sixteen-year trends in overall refraction and age of myopia onset among Chinese children, with a focus on ages 4-6 years. J Glob Health. 2023 Nov 9;13:04144. doi: 10.7189/jogh.13.04144. PMID 37934967
- [Result] Pan Z, Xian H, Li F, Wang Z, Li Z, Huang Y, Liu W, Li Y, Li F, Wang J, Chen H, Wu Y, Xu Y, Wu G, Zhang Y, He L, Zhang J, Zhang F, Qian X, Zhang X, Zhou L, Feng Y, Li L, He X, Xu X, Yang J, Zhou X, Zhu D, Pan C, Ang M, Saw SM, Zheng Y, He M, Jonas JB, Bressler NM, Cheng CY, Tham YC, Zhang C, Wang YX, Wong TY. Myopia and high myopia trends in Chinese children and adolescents over 25 years: a nationwide study with projections to 2050. Lancet Reg Health West Pac. 2025 Jun 11;59:101577. doi: 10.1016/j.lanwpc.2025.101577. eCollection 2025 Jun. PMID 40568343
- [Result] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007